CLINICAL TRIAL: NCT02781857
Title: Exhaled Breath Analysis by Secondary Electrospray Ionization - Mass Spectrometry (SESI-MS) in Patients With Lung Cancer
Brief Title: Mass Spectral Fingerprinting in Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr.2015-0607
Record Dates: First submitted 2016-04-26; First posted 2016-05-25 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
Keywords: Exhaled Breath; Mass Spectrometry; Fingerprinting
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 100 patients with lung cancer: * Group A: 70 patients with any type of lung cancer eligible for lung cancer surgery
  * Group B: 30 patients with any type of lung cancer not eligible to surgery (small-cell carcinoma, squamous cell carcinoma, adenocarcinoma, large-cell carcinoma).
  Interventions: Other: No intervention
- 60 controls: 60 controls (group C) matched for age, gender, smoking history.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
To answer the question whether a disease specific profile of breath in patients with lung cancer can be detected by an untargeted metabolomic study using exhaled breath analysis by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed lung cancer based on cytological or histological analysis.
* Group A: any type of lung cancer eligible for surgical resection (up to TNM stage IIIa).
* Group B: any type of lung cancer (small-cell carcinoma, non-small-cell carcinoma) not amenable for surgical resection.
* Group C: matched controls.
* Age between 18 and 85 years at study entry

Exclusion Criteria:

* Another 'active' secondary malignant disease (e.g. breast cancer, colon carcinoma) in group A and B, presence of any active malignant disease in group C (based on personal information).
* Acute inflammatory disease (e.g. common cold) within the last 4 weeks.
* Any other acute lung disease which affects breath measurements
* Acute or chronic hepatic disease.
* Renal failure or renal replacement therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer will be included according to the predefined inclusion and exclusion criteria.
  Matched controls will be recruited from the general population by printed flyers, newspaper advertisements and personal communication.
Sampling Method: Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of volatile organic compounds (VOCs) in the exhaled breath will be analysed using mass spectrometry | 1 day, single measurement
  The primary outcome will be the lung cancer specific mass spectrometric profile of VOCs of exhaled breath analysis (markers of lung cancer in exhaled breath).

SECONDARY OUTCOMES:
Group A: Concentration of volatile organic compounds (VOCs) in the exhaled breath will be analysed using mass spectrometry before and after lung cancer surgery | Group A: 2 measurements on 2 different days; Day 1: 1. measurement (before surgery), Day 2: (6-12 weeks after surgery): 2. measurement
  The acquired profiles of mass spectral VOCs before and after lung cancer surgery will be analysed for significant differences.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof. MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herth J, Schmidt F, Basler S, Sievi NA, Kohler M. Exhaled breath analysis in patients with potentially curative lung cancer undergoing surgery: a longitudinal study. J Breath Res. 2024 May 17;18(3). doi: 10.1088/1752-7163/ad48a9. PMID 38718786